CLINICAL TRIAL: NCT06199661
Title: Feasibility and Efficacy of a High-Intensity Exercise Intervention in Elderly Healthy Controls
Brief Title: High-Intensity Exercise in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: University of San Francisco (Other)
Responsible Party: Principal Investigator, Maria Ivanova, Research Scientist, University of California, Berkeley
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1884
Record Dates: First submitted 2023-12-13; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Functional Fitness; Cognitive Abilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APEX (Experimental): Physical exercise intervention based on high-intensity interval training
  Interventions: Behavioral: APEX

INTERVENTIONS:
Behavioral: APEX — Three phases: warm-up, high-intensity interval training (HIIT) phase, cool-down. A 10-minute warm-up included deep breathing meditation and dynamic joint mobility exercises. Then, a 40-minute strength and balance workout in HIIT format with five different high-intensity (HI) exercises interspersed with five different postural stability recovery exercises. The HI intervals focused on enhancing cardiovascular fitness, muscle strength, and motor performance. The recovery intervals incorporated balance and mobility exercises. The HI exercises lasted 30 seconds for the first three weeks and then increased to 45 seconds in the fourth week while the recovery exercises lasted 60 seconds throughout the entire intervention. The HIIT phase was repeated three times in the 40 minute block. Lastly, a 10-minute cooldown consisting of standing and seated exercises similar to the warm-up.
  Other Names: Physical exercise intervention incorporating high-intensity interval training

SUMMARY:
The goal of this interventional study was to test the high-intensity interval training called Aphasia Physical Exercise (APEX) in healthy older adults. The main questions it aimed to answer were:

1. what is the safety and feasibility of APEX?
2. what are APEX's acute physiological effects?
3. what is APEX's effects on functional fitness?
4. what is APEX's effects on cognition?

Participants underwent:

* Baseline testing session (#1) with cognitive measures only (a week before the Pre-exercise session);
* Pre-exercise session (#2) with maximum oxygen consumption and heart rate assessment, functional fitness and cognitive measures (3-7 days before the start of the exercise program);
* APEX program, two APEX classes per week for four weeks (eight classes in total);
* Post-exercise session (#3), functional fitness and cognitive measures, (0-2 days after the end of the exercise program).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 50 and 80
* Ambulatory and community-dwelling
* Able to travel to University of San Francisco for weekly exercise classes
* No serious underlying health or neurological conditions

Exclusion Criteria:

* Inability to complete physical function assessment or inability to do a chair stand without using hands
* Use of antidiabetic medications
* Use of testosterone supplement or replacement
* Clinical disorder precluding/interfering with participation or assessments (identified by Physical Activity Readiness Questionnaire (PAR-Q+)), including: unstable angina, arrhythmia, uncontrolled hypertension, end stage renal disease on hemodialysis, lower extremity amputation or paralysis, neurological conditions causing functional or pronounced cognitive impairments, active malignancy except for non-melanomatous skin cancers
* Previous neurological history such as stroke, traumatic brain injury, multiple sclerosis, long-term pre-stroke seizures, Parkinson's, Alzheimer's, etc.
* Unable to provide consent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Attendance Rate | 4 weeks during intervention
  The number of classes attended out of eight total classes.
Heart Rate | 4 weeks during intervention
  Heart rate measured in beats per minute.
Functional Reach Test Distance | Once 3-7 days before start of intervention and once 0-2 days after end of intervention
  The distance in inches of an individual's forward reach with one arm while maintaining a standing position with feet flat on the floor at hip width.
Timed Up-And-Go Time | Once 3-7 days before start of intervention and once 0-2 days after end of intervention
  The number of seconds for an individual to rise from a seated position, walk eight feet, turn around, and return to a seated position.
Number of Steps in 2-minute Step Test | Once 3-7 days before start of intervention and once 0-2 days after end of intervention
  The number of right knee raises completed in two minutes while marching in place and raising each knee to a point midway between the patella (kneecap) and iliac crest (top hip bone).
Number of Repetitions in 30-Second Chair Stand Test | Once 3-7 days before start of intervention and once 0-2 days after end of intervention
  The number of sit-to-stands completed in 30 seconds on a standard 17" seat-height chair with arms folded across the chest.
Visual Search Task Accuracy | Once 10-14 days before start of intervention, once 3-7 days before start of intervention, and once 0-2 days after end of intervention
  Number of correct trials
Visual Search Task Reaction Time | Once 10-14 days before start of intervention, once 3-7 days before start of intervention, and once 0-2 days after end of intervention
  Reaction time on correct trials in seconds
Forward Digit Span | Once 10-14 days before start of intervention, once 3-7 days before start of intervention, and once 0-2 days after end of intervention
  The length of the longest sequence of random digits that a participant can correctly recall twice.
Backward Digit Span | Once 10-14 days before start of intervention, once 3-7 days before start of intervention, and once 0-2 days after end of intervention
  The length of the longest sequence of random digits that a participant can correctly report backward twice.
Forward Spatial Span | Once 10-14 days before start of intervention, once 3-7 days before start of intervention, and once 0-2 days after end of intervention
  The length of the longest sequence of random positions that a participant can correctly recall.
Backward Spatial Span | Once 10-14 days before start of intervention, once 3-7 days before start of intervention, and once 0-2 days after end of intervention
  The length of the longest sequence of random positions that a participant can correctly report backward.
Go/No-Go Task Hits | Once 10-14 days before start of intervention, once 3-7 days before start of intervention, and once 0-2 days after end of intervention
  Hits are the proportion of correct responses on trials when "go" is presented.
Go/No-Go Task Reaction Times | Once 10-14 days before start of intervention, once 3-7 days before start of intervention, and once 0-2 days after end of intervention
  Reaction times are for hit trials only (correct responses when "go" is presented) in seconds.
Flanker Task Accuracy | Once 10-14 days before start of intervention, once 3-7 days before start of intervention, and once 0-2 days after end of intervention
  Number of correct trials.
Flanker Task Reaction Times | Once 10-14 days before start of intervention, once 3-7 days before start of intervention, and once 0-2 days after end of intervention
  Reaction time on correct trials in seconds.
Stroop Task Accuracy | Once 10-14 days before start of intervention, once 3-7 days before start of intervention, and once 0-2 days after end of intervention
  Number of correct trials.
Stroop Task Reaction Times | Once 10-14 days before start of intervention, once 3-7 days before start of intervention, and once 0-2 days after end of intervention
  Reaction time on correct trials in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- University of San Francisco, San Francisco, California, United States